CLINICAL TRIAL: NCT01582412
Title: A Phase 1, Open-Label, Sequential Study of the Effect of Multiple Doses of Isavuconazole on the Pharmacokinetics of a Single Dose of Digoxin in Healthy Adult Subjects
Brief Title: Drug Interaction Study of Isavuconazole and Digoxin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Collaborators: Basilea Pharmaceutica International Ltd (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 9766-CL-0025
Record Dates: First submitted 2012-04-19; First posted 2012-04-20 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Pharmacokinetics of Isavuconazole; Pharmacokinetics of Digoxin; Healthy Volunteers
Keywords: Isavuconazole; Digoxin; Healthy Volunteers; BAL8557
MeSH Terms: interventions — isavuconazole; Digoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Isavuconazole and digoxin (Experimental): Isavuconazole three times per day (TID) on Days 15 and 16, and once daily (QD) on Days 17 thru 26. Digoxin single dose on Days 1 and 19.
  Interventions: Drug: Isavuconazole; Drug: digoxin

INTERVENTIONS:
Drug: Isavuconazole — oral
  Other Names: BAL8557
Drug: digoxin — oral
  Other Names: Lanoxin®

SUMMARY:
The purpose of this study is to assess the effect of multiple doses of isavuconazole on the pharmacokinetics of a single dose of digoxin in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* The subject has a body weight of at least 45 kg and has a body mass index (BMI) of 18.0 to 32.0 kg/m2, inclusive
* Results for aspartate aminotransferase (AST) and alanine aminotransferase (ALT) must be ≤ upper limit of normal and total bilirubin must be ≤ 1.5 mg/dL
* The female subject agrees to sexual abstinence, or is surgically sterile, postmenopausal (defined as at least 2 years at Screening without menses), or using a medically acceptable double barrier method (e.g. spermicide and diaphragm, or spermicide and condom) to prevent pregnancy and agrees to continue using this method from Screening until 3 weeks after the follow-up visit at the end of the study; and is not lactating or pregnant as documented by negative pregnancy tests at Screening and Day -1
* The male subject agrees to sexual abstinence, is surgically sterile, or is using a medically acceptable method to prevent pregnancy and agrees to continue using this method from Screening until 3 weeks after the follow-up visit at the end of the study

Exclusion Criteria:

* The subject has a history of unexplained syncope, cardiac arrest, unexplained cardiac arrhythmia or torsade de pointes, structural heart disease, or family history of Long QT syndrome (suggested by sudden death of a close relative at a young age due to possible or probable cardiac causes)
* The subject has a positive result for hepatitis C antibodies or hepatitis B surface antigen at Screening or is known to be positive for human immunodeficiency virus (HIV)
* The subject has a known or suspected allergy to any of the components of the trial products including digoxin or the azole class of compounds, or a history of multiple and/or severe allergies to drugs or foods (as judged by the investigator), or a history of severe anaphylactic reactions
* The subject is a smoker (any use of tobacco or nicotine containing products) within 6 months prior to Screening
* The subject has had treatment with prescription drugs or complementary and alternative medicines within 14 days prior to Day -1, or over-the-counter medications within 1 week prior to Day -1, with the exception of acetaminophen up to 2 g/day
* The subject has a recent history (within the last 2 years) of drug or alcohol abuse, as defined by the investigator, or a positive drug and/or alcohol screen

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-03; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic (PK) profile for digoxin (in plasma):AUCinf, AUClast, Cmax | Days 1 and 19
  Area under the concentration-time curve (AUC) from time 0 extrapolated to infinity (AUCinf), AUC from time of dosing to the last quantifiable concentration (AUClast), and maximum concentration(Cmax)

SECONDARY OUTCOMES:
PK profile for digoxin (in plasma): tmax, Vz/F, CL/F, and t1/2 | Days 1 and 19
  Time to attain Cmax(tmax), apparent volume of distribution (Vz/F), apparent body clearance after oral dosing (CL/F), and apparent terminal elimination half-life (t1/2)
PK Isavuconazole (in plasma): trough concentration (Ctrough) | Day 17 and Days 21 through 27
PK profile for Isavuconazole (in plasma): AUCtau, Cmax, and tmax | Days 18 and 19
  AUC during time interval between consecutive dosing (AUCtau), maximum concentration (Cmax),and time to attain Cmax (tmax)
Safety assessed by recording of adverse events, clinical laboratory evaluation, electrocardiograms (ECGs) and vital signs. | Day 1 through Day 34 (± 2 days)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development
Locations (1):
- Parexel International, Baltimore, Maryland, United States